CLINICAL TRIAL: NCT01286337
Title: Axillary Lymphadenectomy. A Randomized Trial Comparing Bipolar Vessel Sealing To Conventional Technique
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Gianotti Luca, Milano-Bicocca university
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ligasure; ligamonza
Record Dates: First submitted 2011-01-19; First posted 2011-01-31 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2010-08

CONDITIONS: Axilla Node Dissection
Keywords: axilla; surgery; technique; bipolar vessel sealing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- vessel sealing (Experimental): axilla dissection using this device
  Interventions: Procedure: bipolar vessel sealing
- control (Active Comparator): standard surgical technique
  Interventions: Procedure: control

INTERVENTIONS:
Procedure: bipolar vessel sealing
  Arms: vessel sealing
Procedure: control
  Arms: control

SUMMARY:
lymphorrehea remains the most frequent complication after axillary lymphadenectomy. we hyphothesize that the use of a bipolar vessel sealing may reduce the rate of lymph collection compared to the traditional surgical technique

ELIGIBILITY:
Inclusion Criteria:

* Women with documented breast cancer (by histology or cytology) and candidate to elective axillary lymphadenectomy

Exclusion Criteria:

* Age less than 18 years
* Denied written informed content
* Previous axillary operations (except for sentinel node biopsy)
* Preoperative radio-chemotherapy
* Scheduled reconstructive breast operation

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
reduction of lymphorrhea rate | forth postoperative day

SECONDARY OUTCOMES:
reduction of lymph output from the axillary drain | forth postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: angelo nespoli, md, Study Director — milano-bicocca university; luca gianotti, md, Principal Investigator — milano-bicocca university
Locations (1):
- San Gerardo Hospital, Monza, Italy

REFERENCES:
- [Derived] Nespoli L, Antolini L, Stucchi C, Nespoli A, Valsecchi MG, Gianotti L. Axillary lymphadenectomy for breast cancer. A randomized controlled trial comparing a bipolar vessel sealing system to the conventional technique. Breast. 2012 Dec;21(6):739-45. doi: 10.1016/j.breast.2012.08.003. Epub 2012 Sep 7. PMID 22959311